CLINICAL TRIAL: NCT01481389
Title: The Effect of Theobromine on Blood Lipid Parameters in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10022V
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Cardiovascular Diseases
Keywords: Blood lipids; risk factor for cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Theobromine; Chocolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Theobromine drink (Active Comparator)
  Interventions: Dietary Supplement: Theobromine
- Cocoa drink (Active Comparator)
  Interventions: Dietary Supplement: Cocoa
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Cocoa and theobromine drink (Active Comparator)
  Interventions: Dietary Supplement: Cocoa and theobromine

INTERVENTIONS:
Dietary Supplement: Theobromine — 200 ml drink with added theobromine (no cocoa added)
  Arms: Theobromine drink
Dietary Supplement: Cocoa — 200 ml drink with cocoa (no theobromine added)
  Arms: Cocoa drink
Dietary Supplement: Cocoa and theobromine — 200 ml drink with added cocoa and theobromine
  Arms: Cocoa and theobromine drink
Dietary Supplement: Placebo — 200 ml drink (no added theobromine or cocoa)
  Arms: Placebo drink

SUMMARY:
The purpose of this study is to determine the effect of theobromine on blood lipid parameters in healthy subjects. Secondary objectives are to determine the effect of cocoa and an interaction effect of cocoa and theobromine on blood lipid parameters.

Hypothesis: theobromine has a positive effect on blood lipid parameters.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and post-menopausal women: no medical conditions which might affect study measurements (judged by study physician)
* Willing and able to participate in the study protocol
* Written informed consent
* Age 40-70 years
* 10-year risk of developing CHD <10%, based on data from the Framingham Heart Study
* BMI > 18 and < 30 kg/m2
* Blood pressure, heart rate, haematological and clinical chemical parameters within the normal reference range as judged by research physician
* Willing to comply with the dietary restrictions of the study.
* Accessible veins on arm(s) as determined by examination at screening

Exclusion Criteria:

* Previous cardiovascular event(s) (stroke, TIA, angina, myocardial infarction, heart failure)
* Diabetes mellitus
* Reported alcohol consumption > 14 units/week (female) or > 21 units/week (male)
* Currently on a medically prescribed diet, or slimming diet
* Reported weight loss or gain of 10% body weight or more during a period of 6 months before pre-study examination
* Reported intense sporting activities > 10 h/w
* Use of prescribed medication which may interfere with study measurements, as judged by the physician
* Use of antibiotics in the three months before screening or during the study.
* Currently smoking or being a non-smoker for less than 6 months and reported use of any nicotine containing products in the 6 months preceding the study and during the study itself
* Reported intolerance to test products or other food products provided during the study
* Blood donation 1 month (males) or 2 months (females) prior to screening and during the study
* Reported participation in another nutritional or biomedical trial 3 months before screening or during the study.
* Extreme coffee consumption

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Blood lipids | after 4 weeks intervention

SECONDARY OUTCOMES:
Blood pressure | After 4 weeks intervention
Heart rate | After 4 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wieneke Koppenol, MSc, Study Director — Unilever R&D; Nicole Neufingerl, MSc, Study Director — Unilever R&D
Locations (1):
- Eurofins Optimed, Gières, France

REFERENCES:
- [Derived] Neufingerl N, Zebregs YE, Schuring EA, Trautwein EA. Effect of cocoa and theobromine consumption on serum HDL-cholesterol concentrations: a randomized controlled trial. Am J Clin Nutr. 2013 Jun;97(6):1201-9. doi: 10.3945/ajcn.112.047373. Epub 2013 Apr 17. PMID 23595874